CLINICAL TRIAL: NCT00701025
Title: Mechanisms of Exercise-induced Bronchospasm
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jonathan Parsons, Professor of Clinical Internal Medicine, Ohio State University
Other Study IDs: 2007H0189
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Exercise-induced Bronchospasm
Keywords: inflammation in asthmatic and non-asthmatic participants
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, sputum, urine for pregnancy testing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: 35 asthmatic participants with EIB
- 2: 35 without EIB

SUMMARY:
The term exercise-induced bronchospasm (EIB) describes acute, transient airway narrowing that occurs during, and most often after, exercise. Manifestations of EIB can range from mild impairment of performance to severe bronchospasm and respiratory failure.

The pathogenesis of EIB remains controversial and the role of airway inflammation has not yet been definitively characterized. We plan on comparing markers of inflammation in asthmatic participants with and without EIB at baseline and after bronchoprovocation with eucapnic voluntary hyperventilation testing (EVH). We also will collect demographic information as well as information about asthma control and exercise habits.

DETAILED DESCRIPTION:
At Visit 1, participants will complete questionnaires about demographics, asthma control (if asthmatic) and exercise habits. The participants will have baseline spirometry performed, and skin prick testing for allergies. Skin testing is important as it can influence the level of exhaled nitric oxide and hence we would like to adjust our results for the presence of allergies. Subsequently, volunteers will undergo sputum induction and then have peripheral blood drawn for microRNA analysis. MicroRNA's are single-stranded RNA molecules of about 21-23 nucleotides in length regulating gene expression. Patterns of MicroRNA expression have been linked to heart disease and cancer. Similar patterns have not been identified in exercise-induced asthma. In total, including time for questions and recovery, the time for Visit 1 will be approximately 3 hours.

At Visit 2, which will occur 24 hours to 7 days after Visit 1 in order to minimize risk of asthma exacerbation, the participants will again have baseline spirometry. Baseline exhaled nitric oxide will be performed. Eucapnic Voluntary hyperventilation testing will then be performed. They then will have a second exhaled nitric oxide quantification, will undergo sputum induction and then have peripheral blood drawn for microRNA analysis, all occurring after EVH testing. In total, including time for questions and recovery, the time for Visit 2 will be approximately 2 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. History of physician-diagnosed asthma
3. Age between 18 and 70 years old.
4. Females of childbearing age may participate only if they have a negative pregnancy test, are non-lactating, and agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study. These requirements for contraception also apply to women who may have irregular or absent menstrual periods.
5. Non-smoker for 6 months or longer
6. Less than 10 pack year (number of packs per day (x) years of smoking = pack years) smoking history

Exclusion Criteria:

1. Objective evidence of severe lung impairment on pulmonary function testing performed at the beginning of the study.
2. Participation in another interventional research trial
3. Unable to provide consent
4. Pregnancy
5. Asthma exacerbation within the last 4 weeks.
6. History of severe reaction to allergy skin testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: EIB is one of the most common triggers of bronchospasm in asthmatics. It is identified as a trigger in 80-90% of asthmatics. It also occurs frequently (10-15%) in healthy volunteers without asthma. Inclusion of a heterogenous population of asthmatics and non-asthmatics will help provide much needed information to help compare/contrast EIB that occurs in these two groups.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To compare markers of inflammation in asthmatic participants with and without EIB at baseline and after bronchoprovocation with eucapnic voluntary hyperventilation testing (EVH). | 1 week

SECONDARY OUTCOMES:
to identify important differences between non-asthmatics and asthmatics that suffer from EIB | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P. Parsons, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States